CLINICAL TRIAL: NCT06898385
Title: A Phase I Clinical Study of IX001 TCR-T Injection in the Treatment of Advanced Pancreatic Cancer Patients With KRAS G12V Mutation
Acronym: IX001 TCR-T
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: ImmuXell Biotech Ltd. (Unknown)
Responsible Party: Principal Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IX001 TCR-T
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: IX001 TCR-T injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IX001 TCR-T injection (Experimental): IX001 TCR-T injection targeted for KRAS mutation
  Interventions: Biological: IX001 TCR-T injection; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: IX001 TCR-T injection — IX001 TCR-T injection will be administered intravenously after lymphodepletion.
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
  Other Names: Endoxan

SUMMARY:
This is a single-arm, open-label clinical study to evaluate the safety, tolerability and preliminary efficacy of IX001 TCR-T injection in advanced pancreatic cancer patients with KRAS G12V mutation.

DETAILED DESCRIPTION:
This study will enroll participants with advanced pancreatic cancer patients with KRAS G12V mutation. The study consists of screening period, leukapheresis period, lymphodepletion period, treatment period, observation period and follow-up period. A total of 9-12 evaluable patients are planned to be recruited. The study is planned to be conducted using the "3 + 3" dose escalation design in two dose groups, and a single dose of the study drug will be administered at the dose levels of 3 × 10^9 ± 30% cells and 1 × 10^10 ± 30% cells. Subjects will be enrolled sequentially and treated by IX001 TCR-T injection at the corresponding planned dose level. All subjects who have received IX001 TCR-T injection will be followed for safety and efficacy up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary signing of an informed consent form (for Human Leukocyte Antigen (HLA) typing and tumor gene mutation test, and main screening)
* 2. Males or females, aged 18-75 years (inclusive)
* 3. Patients with pathologically (histopathologically) or cytologically confirmed pancreatic ductal adenocarcinoma
* 4. Patients with unresectable locally advanced or metastatic disease who fail standard of care, i.e., patients who have progression after prior gemcitabine-containing chemotherapy or FOLFIRINOX (oxaliplatin + irinotecan + calcium folinate + 5-FU) or NALIRIFOX (irinotecan liposome + oxaliplatin + calcium folinate + 5-FU) regimen, including those who have progression within 6 months after the end of neoadjuvant/adjuvant therapy
* 5. At least one measurable lesion (according to RECIST 1.1 criteria), specifically: longest diameter of ≥10 mm for non lymph node lesions or shortest diameter of ≥15 mm for lymph node lesions (tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable, unless unequivocal progression of the lesion is demonstrated by an evidence)
* 6. Patients with tumor tissue or peripheral blood tested positive for KRAS-G12V mutation and expression of matching HLA-A*11:01 subtype
* 7. Eastern Cooperative Oncology Group (ECOG) ≤ 1
* 8. Life expectancy ≥3 months
* 9. Adequate functional reserve of organs: A) Hematology requirements (no blood transfusion or hematopoietic stimulating factor treatment within 14 days): Absolute neutrophil count ≥ 1.5×10^9/L; Platelet count ≥ 75×10^9/L, hemoglobin > 90 g/dL; Absolute lymphocyte count ≥ 0.5×10^9/L; B) Blood Biochemistry Requirements: Alanine aminotransferase ≤ 3 × upper limit of normal（ULN） (≤ 5 × ULN for patients with liver metastases); Aspartate aminotransferase ≤ 3 × ULN (≤ 5 × ULN for patients with liver metastases); Creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min; Serum total bilirubin ≤ 1.5 × ULN; C) Coagulation requirements: Partial thromboplastin activity time (APTT) ≤ 1.5 × ULN; International normalized ratio (INR) ≤1.5 × ULN; D) Left ventricular ejection fraction (LVEF) ≥ 50% and no clinically significant pericardial effusion as diagnosed by echocardiography; E) No clinically significant electrocardiographic abnormality; F) Basic oxygen saturation is >92% under the indoor natural air environment.
* 10. Women of childbearing age must be negative for blood Human Chorionic Gonadotropin (HCG) pregnancy test (by immunofluorescence method) at screening and baseline periods, and agree to use effective contraception for at least 1 year after infusion; and male subjects whose partners are women of childbearing age must agree to use effective barrier contraception methods and avoid sperm donation for at least 1 year after infusion.

Exclusion Criteria:

* 1. The subject is currently suffered from or have suffered from other incurable malignant tumors within previous 5 years, except in skin basal cell cancer、carcinoma in situ or breast cancer have received curative treatment with no recurrence within the past 3 years)
* 2. History of organ transplantation
* 3. A history of mental disorders, which may affect compliance with this protocol or lead to failure in signing the Informed Consent Forms(ICF)
* 4. A history of autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis and systemic lupus erythematosus) requiring systemic immunosuppressive/systemic disease-modulating drugs
* 5. Poorly controlled hypertension with drug (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg) or occurrence of grade III-IV heart failure or myocardial infarction, cardiac angioplasty or stent placement, unstable angina pectoris, or other clinically significant heart diseases within one year prior to signing the ICF; QTc interval >450 ms for males or QTc interval >470 ms for females during screening (QTc interval calculated using the Fridericia formula)
* 6. Symptomatic intracranial metastases
* 7. Subjects have ascites or pleural effusion requiring drainage to relieve symptoms or have received drainage within 2 weeks. Asymptomatic participants with a small amount of pleural effusion or ascites on imaging are allowed
* 8. Subjects who have experienced tumor-related intestinal or bowel obstruction within 6 months. including incomplete obstruction related to underlying disease or symptoms of intestinal obstruction requiring treatment
* 9. A history of or any central nervous system disorders, such as epileptic seizure, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system within the past 6 months
* 10. A positive result obtained in any of the following virological tests: A) Antibody to human immunodeficiency virus (HIV antibody); B) Hepatitis C virus antibody (HCV antibody), with a positive result for hepatitis C virus ribonucleic acid (HCV RNA); C) Positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA) copies ≥2000 IU/mL; D) Treponema pallidum antibody (TP antibody) and positive for unheated serum reagin test;
* 11. Fungal, bacterial, viral or other infections or suspected fungal, bacterial, viral or other infections that cannot be controlled or require intravenous administration
* 12. Significant tendency for bleeding, such as active gastrointestinal bleeding, coagulation disorders
* 13. Deep vein thrombosis requiring treatment within the past 6 months, unless the risk of thrombosis is acceptable after treatment, as assessed by the investigator
* 14. Interstitial lung disease (such as interstitial pneumonia, pulmonary fibrosis), or a history of clinically significant respiratory system diseases at screening
* 15. Use of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks prior to leukapheresis
* 16. Receipt of gene therapy or other cell therapies within the past 6 months
* 17. Participation in any other clinical studies within 28 days prior to signing the master informed consent form, or the date of signing the master informed consent form still within 5 half-lives of the drug from the last dose in the last clinical study (whichever is longer)
* 18. Patients with poor compliance due to physiological, family, social, geographic and other factors, and failure to follow the study protocol and the follow-up plan
* 19. Patients with contraindications to drugs used in the study
* 20. Comorbidities requiring treatment with systemic corticosteroids (dexamethasone at a dose of ≥ 5 mg/day or other corticosteroids at the equivalent dose) or other immunosuppressive drugs after initiation of the study treatment, as judged by the investigator
* 21. Women who are breastfeeding and are unwilling to stop breastfeeding
* 22. Any other conditions that are, in the opinion of the investigator, not suitable for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-03-27 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | 4 weeks
  Proportion of patients with DLT
Adverse Events (AEs) | 2 years
  Incidence and severity of adverse events
Serious Adverse Events (SAEs) | 2 years
  Incidence and severity of serious adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1
Disease Control Rate (DCR) | 2 years
  The percentage of participants who achieved Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1
Changes in Serum Tumor Markers compared to Baseline | 2 years
  Changes of tumor markers in serum detected by immunofluorescence compared to baseline level, including carbohydrate antigen 19-9 (CA19-9), carcinoembryonic antigen (CEA), and carbohydrate antigen 12-5 (CA12-5)
Duration of response (DOR) | 2 years
  DOR is defined as the time from the first evaluation of a tumor as CR or PR to the first evaluation as progressive disease (PD) or death from any cause
Time to response (TTR) | 2 years
  TTR is defined as the time between cell infusion and initial disease assessment as CR or PR
Progression-free survival (PFS) | 2 years
  PFS is defined as the time from the date of cell infusion until the date of tumor progression or death from any cause
Overall survival (OS) | 2 years
  OS is defined as the time between the date of cell infusion and the death of the patient for any reason
TCR gene copies | 2 years
  TCR gene copies detected by quantitative polymerase chain reaction (qPCR) in peripheral blood
TCR-T cell counts | 2 years
  TCR-T cell counts detected by flow cytometry in peripheral blood
Pharmacodynamic of IX001 TCR-T injection | 2 years
  Peak TCR-T cell count (Cmax), Time to peak (Tmax) ,Area under the peripheral blood concentration versus time curve (AUC)
Changes in cytokine level | 2 years
  Calculate the change of cytokine level in peripheral blood after IX001 TCR-T injection infusion. Cytokines include interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α), and interferon-gamma (IFN-γ), etc
Changes in lymphocyte subpopulations | 2 years
  Calculate the change of lymphocyte subpopulations in peripheral blood by flow cytometry after IX001 TCR-T injection infusion. lymphocyte subpopulations include CD3+T cell, CD4+T cell,CD8+T cell, etc
Proportion of patients with anti-IX001 antibodies | 2 years
  Anti-IX001 TCR-T injection Antibodies in peripheral blood after IX001 TCR-T injection infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided